CLINICAL TRIAL: NCT00702832
Title: Effects of Vestibular Rehabilitation in the Treatment of Patients With Acute Vestibular Loss. - A Randomized Controlled Trial
Brief Title: Effect of Vestibular Rehabilitation - a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Haukeland University Hospital (Other); St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REK 4.2007.1802
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Dizziness; Nausea; Nystagmus; Vestibular Diseases
Keywords: Vestibular rehabilitation; acute vestibular injury; Dizziness; Nausea; Nystagmus; Daily life activities; Balance; physiotherapy
MeSH Terms: conditions — Dizziness; Nausea; Nystagmus, Pathologic; Vestibular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular rehabilitation (Experimental): early supported vestibular rehabilitation
  Interventions: Behavioral: Vestibular rehabilitation
- standard (Active Comparator): standard treatment
  Interventions: Other: standard treatment

INTERVENTIONS:
Behavioral: Vestibular rehabilitation — Daily home training (4-6 specific exercises) 2-3 times per day. Group training led by a physiotherapist twice per week during the first 10 weeks and once per week from 10 weeks to 12 months or to symptoms are cured.
  Arms: Vestibular rehabilitation
Other: standard treatment — treatment as usual
  Arms: standard

SUMMARY:
The aim of this study is to assess if early supported vestibular rehabilitation can reduce dizziness and improve daily life activities in patients with acute vestibular injury.

The study question is: Does early supported vestibular rehabilitation have an additional effect on dizziness symptoms and daily life functions compared to standard treatment?

ELIGIBILITY:
Inclusion Criteria:

* acute symptoms of dizziness, nausea and nystagmus
* diagnosed by videonystagmography (at least 25% reduced caloric response in one ear)
* age 18-70 years
* inclusion within one week after symptom debut

Exclusion Criteria:

* chronic dizziness
* psychiatric diagnosis that might interfere with participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
vertigo | at inclusion, 10-12 weeks, 12 months
  Vertigo symptom scale (VSS)

SECONDARY OUTCOMES:
Dizziness | At inclusion, 10-12 weeks, 12 months
  Dizziness Handicap Inventory (DHI), University of California Los Angeles Dizziness Questionnaire (UCLA-DQ), Three questions regarding dizziness on VAS-scale,
Movement provoked dizziness | at inclusion, 10-12 weeks, 12 months
  Rombergs test and advanced Rombergs test
return of symptoms | 12 months
sick leave | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Siv Mørkved, PhD, Principal Investigator — Associate professor / senior researcher
Locations (1):
- St. Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Tokle G, Morkved S, Brathen G, Goplen FK, Salvesen O, Arnesen H, Holmeslet B, Nordahl SHG, Wilhelmsen KT. Efficacy of Vestibular Rehabilitation Following Acute Vestibular Neuritis: A Randomized Controlled Trial. Otol Neurotol. 2020 Jan;41(1):78-85. doi: 10.1097/MAO.0000000000002443. PMID 31789800